CLINICAL TRIAL: NCT02669771
Title: Xtandi® Capsules 40 mg Protocol for Long-Term Specified Drug Use-Results Survey
Brief Title: Long-Term Specified Drug Use-Results Survey for Xtandi Capsule
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 9785-MA-1018
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Xtandi; MDV3100; long term use; enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enzalutamide group: oral
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: Xtandi; MDV3100

SUMMARY:
The purpose of this study is to confirm the long term safety and efficacy of enzalutamide in patients.

ELIGIBILITY:
Inclusion Criteria:

* no history of treatment with enzalutamide

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with castration-resistant prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Incidences of Adverse Events | Up to 2 years

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years
Change from baseline in PSA value | Up to 2 years
  PSA: prostate-specific antigen

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Numakunai, Iwate
  - Aichi
  - Akita
  - Aomori
  - Chiba
  - Ehime
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Gunma
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Ishikawa
  - Kagawa
  - Kagoshima
  - Kanagawa
  - Kochi
  - Kumamoto
  - Kyoto
  - Mie
  - Miyagi
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nara
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shiga
  - Shimane
  - Shizuoka
  - Tochigi
  - Tokushima
  - Tokyo
  - Tottori
  - Toyama
  - Wakayama
  - Yamagata
  - Yamaguchi
  - Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.